CLINICAL TRIAL: NCT07333768
Title: EQUISOCK: New Antiequine for Ankle
Brief Title: EQUISOCK: New Antiequine
Acronym: EQUISOCK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Rocío Llamas-Ramos, Principal Investigator, University of Salamanca
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Device Feasibility
Other Study IDs: EQUISOCK2026; University of Salamanca (Other Grant/Funding Number: University of Salamanca)
Record Dates: First submitted 2025-12-08; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Ankle (Ligaments); Instability (Old Injury); Ankle Equinus; Ankle Dorsiflexion

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EQUISOCK group (Experimental): Participants must wear the new ankle orthosis during assessments and in their daily lives for at least one month, which is the duration of the study.
  Interventions: Device: EQUISOCK
- Other ankle orthosis (Active Comparator): Participants must wear the conventional ankle orthosis (and without orthosis) during assessments and in their daily lives, before wear the new one.
  Interventions: Device: Other ankle orthosis

INTERVENTIONS:
Device: EQUISOCK — Participants must wear the new ankle orthosis during assessments and in their daily lives for at least one month, which is the duration of the study.
  Arms: EQUISOCK group
Device: Other ankle orthosis — Participants must wear the conventional ankle orthosis and without orthosis, during assessments and before wearing the new one
  Arms: Other ankle orthosis

SUMMARY:
The goal of this experimental study is to test the feasibility and validity of a new orthosis in patients with ankle lesions (external popliteal sciatic nerve or nerve injuries resulting in loss of ankle dorsiflexion) of both sexes and all ages. The main question it aims to answer is:Is the new orthosis a support for ankle stability??Does the new orthosis improve ankle function and patients' quality of life??The control group will be the subjects themselves when wearing their conventional ankle orthosis or without it. Participants must wear the new ankle orthosis for at least one month to assess the effectiveness of the orthosis and evaluate any changes that have occurred in the ankle joint and muscles.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic ankle injuries
* patients with external popliteal sciatic nerve lesion or nerve injuries resulting in loss of ankle dorsiflexion
* patients who have already been prescribed an orthosis
* patients of all ages

Exclusion Criteria:

* inability to stand actively and stably
* inability to walk unaided
* inability to follow instructions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Device Feasibility | Baseline and up to 4 weeks
  Device feasibility will be assessed through participants' awareness of the device, as an indicator of its accessibility, visibility, and potential for effective implementation within the target population. A self diary Will be requested

SECONDARY OUTCOMES:
Ankle function with virtual reality | Baseline and up to 4 weeks
  Ankle function will be assessed using a virtual reality programme that requires movement of the lower limb to assess ankle stability, with and without orthosis. The assessment will be using a Borg scale (range of effort that the individual perceives when exercising). From 0 points (minimum effort) to 10 points (maximum effort).
Range of motion with Gyko device | Baseline and up to 4 weeks
  The range of motion of the knee joint will be measured using the Gyko device with and without the new orthosis. The assessment will be in degrees (from 0 to 120º)
Footprint with a pressure platform | Baseline and up to 4 weeks
  The distribution of static and dynamic load will be assessed with and without orthosis, using a pressure platform, as well as static balance with eyes open and closed and dynamic balance. The assessment will be the percentage of support from the sole of the foot in each movement.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salamanca, Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No